CLINICAL TRIAL: NCT05728437
Title: Effect of Resistance Exercises in Reducing Plasma Liver Enzymes Level Post Burn.
Brief Title: Effect of Resistance Exercises on Liver Enzymes Post Burn.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Gamal Fawzy El-Sayed, Lecturer of physical therapy of surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003633
Record Dates: First submitted 2023-01-19; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): This group includes 30 burned patients who will receive resistance exercises 8 weeks (3times/week) by using dumbbells and sand bags in addition to their physical therapy program (splinting, stretching ex. and ROM ex.) and medical treatment.
  Interventions: Procedure: Resistance exercise
- Control group (No Intervention): This group includes 30 burned patients who will receive their physical therapy program (splinting, stretching ex., strengthening ex. and ROM ex.) and medical treatment.

INTERVENTIONS:
Procedure: Resistance exercise — The program will consist of seven exercises: triceps press, biceps curl, lat pull down, calf raise, leg press, leg extension and sit-ups using dumbbells and sand bags. Each session will last approximately 45 minutes and consist of a 5-minute warm-up with stretching following by resistance exercise that will be done as a cir¬cuit, ending with 5-minute cool down. The 1 repetition maximum (1RM) is measured at baseline and follow¬ing the intervention. Initially, participants will do two circuits using 50% of their 1RM and repeat them 10 times for the first and second weeks, progressing to two circuits, using 60% of their 1RM and repeat 10 times for the third and fourth weeks. In fifth and sixth weeks, participants will do three circuits using 60% of their 1RM and repeat 10 times. In the last two weeks, patients will do three circuits using 70% of their 1RM and repeat 10 times. A 90-second rest will be allowed between sets of exercises.
  Arms: Study group

SUMMARY:
Resistance training will be performed for 8 weeks with thrice-weekly sessions on non-consecutive days. The program will consist of seven exercises: triceps press, biceps curl, lat pull-down, calf raise, leg press, leg extension and sit-ups using dumbbells and sandbags. Each session will last approximately 45 minutes and consist of a 5-minute warm-up with stretching followed by a resistance exercise that will be done as a circuit, ending with a 5-minute cooldown. The 1 repetition maximum (1RM) is measured at baseline and following the intervention. Initially, participants will do two circuits using 50% of their 1RM and repeat them 10 times for the first and second weeks, progressing to two circuits, using 60% of their 1RM and repeating 10 times for the third and fourth weeks. In the fifth and sixth weeks, participants will do three circuits using 60% of their 1RM and repeat 10 times. In the last two weeks, patients will do three circuits using 70% of their 1RM and repeat 10 times. A 90-second rest will be allowed between sets of exercises (Hallsworth et al., 2011).

DETAILED DESCRIPTION:
Sixty patients who have partial thickness burn with burned body surface area (BBSA) about 30% to 50% will participate in this study after their release from intensive care unit. Their ages will be ranged from 20 to 45 years. The participants will be selected from Orabi hospital and randomly distributed into two equal groups.

1. Group A (Study group): This group includes 30 burned patients who will receive resistance exercises 8 weeks (3times/week) by using dumbbells and sand bags in addition to their physical therapy program (splinting, stretching ex. and ROM ex.) and medical treatment.

1. Group B (Control group): This group includes 30 burned patients who will receive their physical therapy program (splinting, stretching ex., strengthening ex. and ROM ex.) and medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* The subject selection will be according to the following criteria:
* Age range between 20-45 years.
* Male and female patients will participate in the study.
* All patients have burn with BBSA about 30% to 50%.
* All patients enrolled to the study will have their informed consent.

Exclusion Criteria:

* The potential participants will be excluded if they meet one of the following criteria:
* Cardiac diseases.
* Burn of sole of foot.
* Exposed hand or foot tendons.
* Lower limb amputation.
* History of liver diseases.
* Body mass index (BMI=kg/cm2)<30%.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-19 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
EFFECT OF RESISTANCE EXERCISE ON LIVER ENZYMES POST BURN. | Two month
  plasma liver enzymes level (AST and ALT enzymes)